CLINICAL TRIAL: NCT07268898
Title: National Multicenter Retrospective Real-World Study on the Treatment Status of Newly Diagnosed and Persistent Primary Immune Thrombocytopenia (ITP) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang Lei, MD, Chief Physician, Institute of Hematology & Blood Diseases Hospital, China
Other Study IDs: QT2025009
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: RWS
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated Group
- Untreated Group

SUMMARY:
This study is a nationwide, multicenter, retrospective, real-world, non-interventional (observational) investigation. It retrospectively collects data on treatment modalities and therapeutic responses in patients with newly diagnosed or persistent immune thrombocytopenia (ITP), documents disease progression in both treated and untreated patients, and records the treatment regimens selected by those receiving therapy. The study aims to observe and evaluate the current treatment landscape for newly diagnosed and persistent ITP patients, while also analyzing the efficacy and safety in the treated population. All patient treatments and disease management are solely based on routine clinical practice and are not influenced by this study.

DETAILED DESCRIPTION:
Currently, there is a lack of data on the treatment landscape for newly diagnosed and persistent ITP in China. No information is available regarding the proportion of treated and untreated patients, treatment choices, or therapeutic outcomes in this population. This study retrospectively collects data on treatment approaches and response outcomes in patients with newly diagnosed or persistent ITP, documenting disease progression in both treated and untreated individuals, as well as the treatment regimens selected by those receiving therapy. It aims to observe and analyze the current treatment patterns for newly diagnosed and persistent ITP patients in China, with the goal of clarifying the treatment needs for thrombopoietin receptor agonists (TPO-RAs) in this population. Additionally, the efficacy and safety of treatments in the studied cohort will be evaluated. This study is designed to observe and assess the current treatment status of patients with newly diagnosed and persistent ITP.

ELIGIBILITY:
Inclusion Criteria:

* Availability of traceable inpatient medical records;

Clinically diagnosed with newly diagnosed or persistent ITP (ITP disease course ≤12 months) between July 2021 and September 2025;

Baseline platelet count <30×10⁹/L;

Age ≥6 years;

Inclusion of patients regardless of ITP treatment status, encompassing those receiving any ITP-directed therapy (excluding emergency treatments such as platelet transfusion) and untreated patients (who have not received ITP-specific treatments including glucocorticoids, intravenous immunoglobulin, TPO-RAs, splenectomy, and rituximab).

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients deemed ineligible for the study based on the investigator's judgment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a platelet count ≥30×10⁹/L within 8 weeks, with at least a twofold increase from baseline, and no bleeding manifestations | 2026.2.25

IPD SHARING:
Plan to Share IPD: No